CLINICAL TRIAL: NCT07127848
Title: Comparing Outcomes in Patients Who Underwent Septoplasty With Mucotomy, Turbinectomy, Or Valvuloplasty
Brief Title: Investingation on Outcomes After Combining Septoplasty With Additional Procedures.
Acronym: NOSEjob
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Andro Košec, MD, PhD, Consultant Otorhinolaryngologist and Head and Neck Surgeon, University Hospital Sestre Milosrdnice
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-001
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Nasal Patency; Breathing Disorder During Sleeping; Breathing Mechanics
Keywords: septoplasty; turbinectomy; Valvuloplasty; mucotomy; breathing outcome; nasal breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into three groups: those undergoing septoplasty with turbinectomy, those undergoing septoplasty with flaring sutures of the internal nasal valve and those undergoing septoplasty with radiofrequent ablation of the inferior nasal turbinates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Septoplasty with Mucotomy (Active Comparator): Septoplasty accompanied by radiofrequent mucotomy of the inferior nasal turbinates.
  Interventions: Procedure: Septoplasty with Valvuloplasty
- Septoplasty and Turbinectomy (Active Comparator): Septoplasty accompanied by surgical resection of the inferior nasal turbinates.
  Interventions: Procedure: Septoplasty with Mucotomy
- Septoplasty and Valvuloplasty (Active Comparator): Septoplasty accompanied by placing a flaring sutture in the internal nasal valve area.
  Interventions: Procedure: Septoplasty with Turbinectomy

INTERVENTIONS:
Procedure: Septoplasty with Mucotomy — Subtotal reconstruction of the nasal septum accompanied by radiofrequent nasal mucosal reduction of the inferior turbinates.
  Arms: Septoplasty and Turbinectomy
Procedure: Septoplasty with Turbinectomy — Subtotal reconstruction of the nasal septum accompanied by surgical resection of the inferior turbinates.
  Arms: Septoplasty and Valvuloplasty
Procedure: Septoplasty with Valvuloplasty — Subtotal reconstruction of the nasal septum accompanied by surgical intervention by placing a flare sutture in the internal nasal valve area.
  Arms: Septoplasty with Mucotomy

SUMMARY:
The aim of this study will be to compare postoperative nasal airflow and symptom improvement using a NOSE form in patients after different types of surgical treatment. Patients will be treated with one of the following operations: septoplasty with turbinectomy, septoplasty with radiofrequent ablation of the nasal turbinates, or septoplasty with valvuloplasty.

This is a single-center prospective randomized interventional comparative study on patients in a tertiary rhinology center, who will undergo septoplasty alongside one additional rhinologic procedure aimed at improving nasal patency.

DETAILED DESCRIPTION:
Inclusion criteria will be met if patients are 18 years and above, without any disease or condition affecting nasal breathing apart from allergic rhinitis, septal deviation, hypertrophy of the nasal turbinates. The criteria require complete follow-up during the testing phases, complete documentation, written informed consent and all questionnaire-related data to be complete.

The patients will be divided into three groups: those undergoing septoplasty with turbinectomy, those undergoing septoplasty with flaring sutures of the internal nasal valve and those undergoing septoplasty with radiofrequent ablation of the inferior nasal turbinates. Randomization will be performed via a binary coin-toss method, with allocation con-cealment, and using a heads-tails method on a true random number generator online service (TRNG).

Patients with a history of psychological or mental illness, prior nasal surgery or nasal polyposis will be excluded from the study. Use of any medication related to airway management or nasal patency, such as decongestants or mucolytics, or nasal dilators to influence the external and internal nasal valve function during the study period was not allowed.

Written informed consent will be obtained from all of the eligible patients. Primary outcome measures include subjective NOSE (Nasal Obstruction Symptom Evaluation) questionnaire scores - internationally validated scale for assessment of intensity of nasal obstruction, consisting of 5 claims related to nasal obstruction divided into Likert scales of 4 points for each claim (normal values 2.75-7, with scores >7 indicating clinically relevant nasal obstruction), and objective peak nasal inspiratory flow measurements using a calibrated instrument (PNIF, GM Instruments, with normal values ranging from 130-140 l/min for healthy young adults), while anthropometric and demographic variables will be covariates[12].

PNIF is a noninvasive, easy to perform method commonly used to assess nasal patency. It is a physiologic measure indicating the peak nasal airflow in liters per minute achieved during maximal forced nasal inspiration [ ]. To reduce test-retest variability and sampling bias due to the influence of the elasticity of the lateral nasal wall (the valve effect), three PNIF measurements will be performed preoperatively and repeated at onset and three months postoperatively, with the best measurement recorded for data analysis.

The study was designed to comply with CONSORT guidelines. A minimal study sample of 90 was calculated based on 80% study power and alpha error rate of 5% (G*Power t-test).

ELIGIBILITY:
Inclusion Criteria:

* Patients were 18 years and above, without any disease or condition affecting nasal breathing apart from allergic rhinitis, septal deviation, hypertrophy of the nasal turbinates.

Exclusion Criteria:

* Patients with a history of psychological or mental illness, prior nasal surgery or nasal polyposis were excluded from the study. Use of any medication related to airway management or nasal patency, such as decongestants or mucolytics, or nasal dilators to influence the external and internal nasal valve function during the study period was not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-09-03 (Estimated)

PRIMARY OUTCOMES:
PNIF | Every months until six months postoperatively.
  Peak Nasal Inspiratory Flow measurement - objective measurement of nasal patency in liters per minute.
NOSE questionnaire | Every month up to 6 months post surgery.
  Validated PROM regarding subjective nasal patency assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Andro Košec, MD, PhD, FEBORL-HNS, FACS, Study Chair — University Hospital Center Sestre milosrdnice, Department of ORL&HNS
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez AK, Uhl C, Haehner A, Cuevas M, Hummel T. Objective nasal airflow measures in relation to subjective nasal obstruction, trigeminal function, and olfaction in patients with chronic rhinosinusitis. Rhinology. 2024 Aug 1;62(4):394-402. doi: 10.4193/Rhin23.270. PMID 38507726